CLINICAL TRIAL: NCT03896139
Title: Identification of PAthways of Kinase Inhibitors TOxicity Through Patient Databases
Brief Title: Identification of PAthways of Kinase Inhibitors TOxicity
Acronym: PAKITO
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Investigator, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-1906
Record Dates: First submitted 2019-03-25; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Kinase Inhibitors Toxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- VUMC EHR cohort: De-identified version of the electronic health record (EHR) at Vanderbilt University Medical Center (VUMC).
  Interventions: Drug: Kinase inhibitor
- Toxicity induced by kinase inhibitors in Vigibase database: Case reported in the World Health Organization (WHO) of toxicity or complication of patient treated by KIs, with a chronology compatible with the drug toxicity
  Interventions: Drug: Kinase inhibitor

INTERVENTIONS:
Drug: Kinase inhibitor — Patients treated with kinase inhibitors for cancer or other conditions

SUMMARY:
The investigators are identifying clinical diagnoses and toxicities associated with kinase inhibitors prescription. This identification will be applied will be applied in an electronic-health-record (EHR) cohort including North American and European.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with a kinase inhibitor
* Patient identified in the VUMC EHR cohort or having a toxicity reported in the VigiBase

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with kinase inhibitors or drugs targeting kinase pathways for a cancer with at least one report accessible in the VUMC electronic health record database and/or in VigiBase, the WHO's international pharmacovigilance database.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the incidence of kinase inhibitor (KIs) induced toxicities in health records and their associations with co-medications to identify new mechanisms of drug induced toxicity | population included in VUMC database and/or WHO's database resource up to march 2019
  Identification of a mechanism of a toxicity associated with a KI using comedications and comparing it to reported outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided